CLINICAL TRIAL: NCT05287828
Title: Retrospective Study for the Validation of an Automatic Software for Geometric Measurements of the Principal Arteries and Calcification Detection on Patients With Aortic Aneurysm.
Brief Title: Validation of a Software and the Follow-up of Anteropoterior Migration of Stent
Acronym: ASMOT
Status: Completed | Type: Observational
Sponsor: Nurea (Industry)
Responsible Party: Sponsor
Other Study IDs: ASMOT
Record Dates: First submitted 2022-03-02; First posted 2022-03-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Aortic Aneurysm
Keywords: Software; Automatic; Aneurysm; Scan; Artificial Intelligence; Automatic segmentation; Automatic EVAR indicators
MeSH Terms: conditions — Aortic Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Indicators validation - Group A: This group is composed with the contrasted pre-op CT scan of the 40 patients recruited.
  The classification criterion is "contrasted CT scan".
  Interventions: Other: Surgeons CT scan analysis; Device: PRAEVAorta CT scan analysis
- Indicators validation - Group B: This group is composed with the non-contrasted CT scan of the 40 patients recruted.
  This group is composed with pre-op non-contrasted CT scans to validate the possibility to use the device on the first scan realised on patient, when there is a suspicion of a disease. The classification criterion is "non-contrasted CT scan".
  Interventions: Other: Surgeons CT scan analysis; Device: PRAEVAorta CT scan analysis
- Indicators validation - Group C: This group is composed with the post-op contrasted CT scan of the 35 pathological patients listed above (25 AAA, 5 TAA, 5 JAA).
  This last group is composed with post-op CT scans. These scans are realised in a purpose of follow-up. The classification criterion is "post-op CT scan of patient with a AAA, TAA or JAA".
  Interventions: Other: Surgeons CT scan analysis; Device: PRAEVAorta CT scan analysis
- Indicators validation - Group D: This group is composed with the post-op non-contrasted CT scan of the 35 pathological patients above (25 AAA, 5 TAA, 5JAA).
  To decrease risks for patients, practicians are doing more non-contrasted CT scan. Moreover, they still need the indicators to realize the follow-up of the patient after its surgery. This group is to evaluate the possibility for the software to analysis this type of scan. The classification criterion is "post-op non-contrasted CT scan of patient with a AAA, TAA or JAA".
  Interventions: Other: Surgeons CT scan analysis; Device: PRAEVAorta CT scan analysis
- Stent migration group: 25 patients are added to the 25 patients treated with EVAR (25 AAA) recruted in part 1 in order to have more significative results.
  Interventions: Device: PRAEVAorta CT scan analysis

INTERVENTIONS:
Other: Surgeons CT scan analysis — Surgeons extract indicators using standard methods of analysis
  Groups: Indicators validation - Group A; Indicators validation - Group B; Indicators validation - Group C; Indicators validation - Group D
Device: PRAEVAorta CT scan analysis — CT scans are analysed using PRAEVAorta Suite which is composed of the software PRAEVAorta 2 and PRAEVAorta Web. Indicators extraction is fully automatic.

SUMMARY:
The treatment of aortic aneurysms is today based on different indicators (diameters, lengths, angles, volumes of the arteries) measured on CT scan images. Several indicators are time consuming and complicatated to measure. They demand training and practice. Nurea is developing a software for automatic measurement of these indicators, PRAEVAorta® 2, to facilitate and assist the physician in his clinical routine. The purpose of this study is to compare the analysis realised by the software PRAEVAorta® 2 with the analysis realised by the healthcare professional on retrospective CT scan images.

Contrasted and non-contrasted, pre-operation or post-operation CT scans from 50 patients will be analysed.

The main objectif is to validate the accuracy of the software by demonstrating its adequacy to the standard method of analysis.

The second objectives are the following:

* Evaluate the security of the software PRAEVAorta® 2
* Evaluate the unanticipated risks related to the use of the software
* Validate the accessory PRAEVAorta® Web

We make the following assumption :

90% of the patients show 90% of adequacy to the healthcare professional analysis

DETAILED DESCRIPTION:
Control and quality assurance will be applied in the investigation site. The monitor mandated by the sponsor Nurea will ensure the follow-up and the proper completion of the study, the collection of data in writing, their documentation, recording and report, in accordance with the procedures in place and in accordance with good clinical practice as well as the laws and regulations in force.

Quality control visits realised at regular intervals will be realised by the monitor. During those visits, the following elements could be demanded:

* Informed consent forms, information note
* Respect of the plan of the study and the procedures defined in it
* Quality of the data collected in the Case Report Form (CRF): accuracy, missing data, consistency of data with the "source" documents (medical file, appointment book, originals of laboratory results).
* Management of any products
* Security data All contacts made will give rise to a specific written report

Three type of visits (quality control) will be realised:

* The initiation visit (realised in person) will concern every person potentially involved in the investigation. This visit will be about presenting the plan, redefine inclusion objectives, recall everyone's responsibility and the regulation, as well as answering question.
* The monitoring visits will be realised by the monitor after the first inclusion to ensure the respect of the plan and the regulation, as well as the quality of the collected data. Those visits will be realised every 2weeks, but the frequency can vary regarding the complexity of the study, of the number and the pace of inclusions. Therefore, there will be at least one visit per month.
* The close-out visit will be realised after the last data have been collected. The purpose of this visit is to verify the quality of the collected data, to update the documents before archiving.

In addition to these on-site travels, a regular monitoring over the phone will be realised in order to best support the participating physicians throughout the study.

These quality controls are supplemented by regular follow-up audits in order to evaluate the quality of collected data and to crop the study. An audit may be conducted at any time by persons appointed by the sponsor and independent of the persons conducting the research. Its purpose is to verify the participants' safety and respect for their rights, compliance with applicable regulations and the reliability of data.

An inspection can also be carried out by a competent authority (ANSM for France or EMA in the context of a European study, for example).

The audit, as well as the inspection, can be applied at all stages of the research, from the development of the protocol to the publication of the results and the classification of the data used or produced as part of the research.

Data management Access to data Only participating physicians and the monitor (or clinical research staff) will have access to source files during the monitoring visits.

During quality control visits, the principal investigator must make the following documents available:

* informed consent,
* briefing notes,
* observation notebooks,
* source documents (medical records, appointment books, etc.) In accordance with the law in force, patients have a right of access to their medical file. According to the law of January 2002, patients will be told where they can inquire about the results of the study.

Guidelines for collecting data The term "Case Report Form (CRF)" designates any document whatever its support (for example paper, optical, magnetic or electronic) intended to collect in writing all the information required by the protocol concerning each person who is suitable for research and to be sent to the sponsor.

All the information required by the protocol must be recorded in case report forms and an explanation must be provided for any missing data. The data will have to be collected as and when they are obtained and transcribed in these notebooks in a clear and legible way.

It is the responsibility of the investigator to complete the CRF, but he may delegate this task to the clinical trial technicians or to the research nurse, provided that he has previously completed a task delegation form.

Data collection will be done using e-CRF that will include patient characteristics and study data. The patient will be identified by an alphanumeric code and the data concerning him/her will be anonymized in the form. The code will be reported on all pages of the observation book.

Modification of e-CRF data Corrections of errors which have occurred in an e-CRF will be carried out via the correction module thereof, and must be dated, initialed, and justified.

The copies of the observation notebooks will be kept for at least 15 years on the investigation site while the original copy, once the quality control has been carried out, will be archived by the sponsor for the same duration.

Standard operating procedures Investigators will determine whether patients meet the inclusion criteria, and whether the use of one or the other device will bring them beneficial results.

Screening / pre-selection The selection of the patients is realised by the principal investigator. A first screening of the patient that could be included in the study is realised.

To be pre-included, those patients shall:

1. respect the selection criteria (inclusion and exclusion criteria),
2. have given their consent form by non-opposition
3. Have been treated and /or followed by the hospital

The discrimination of the group of patients is carried out according to the list above.

Reception of the consent form / inclusion The consent form is obtained by non-opposition. The information note and consent form are sent to the pre-selected patient. After one month without any manifestation (refusal) from the patient, the consent is considered as acquired.

The inclusion is validated when all data (cited above) are registered in the e-CRF.

When the consent of the patient has been received, the following data are registered in the e-CRF:

* Demographic data: age, gender
* Scan references: scan manufacturer, contrasted or not, pre- or post-operation scan, scan date
* Investigation data: Patient number, date of signature of the consent
* Images data: Pre-operation scan, post-operation scan The inclusion is validated when all data (cited above) are registered in the e-CRF.

Sample size assessment

The number of patients needed is calculated to answer the main objective of this study which is the validation of the de vice PRAEVAorta® 2. The study realised on the first version of the medical device PRAEVAorta® has shown a proportion of 93% of patient with measures calculated by the software in adequation with the measures realised following the standard method of analysis (ratio ≥ 90%). Because the new version of the software PRAEVAorta® 2 has been improved, we expect to observe the same proportion.

Patient number calculation:

Hypotheses are the following:

H0: The proportion of patients with an absolute mean discrepancy > 5mm is 90% H1: The proportion of patient with an absolute mean discrepancy ≤ 5mm is strictly over 90% For this statistical analysis, variables are quantitative: aorta measurements. We consider over here the proportion of patients per sub-group who have as less or greater than 90%.

Comparison of two proportions: a theoretical proportion with an observed proportion The theoretical proportion ϕ0 is 90%

n=([1,96(φ0(1-φ0))^0,5 +u2β(φ(1-φ))^0,5]^2)/([φ0-φ]^2)=32

For security reasons and to anticipate any problem we choose to include approximately 25% more subjects. Therefore, the total of patient is 40. We add 15 additional patients to meet the ancillary objective of evaluating anteroposterior migration of stents. The total is then 65 patients.

Patients will be devided in 4 groups related to the type of scan analysed

Images' analysis Pseudonymised pre-operation and post-operation thin-sliced CT images in DICOM format will be analysed.

This study is design in two parts:

Part 1: Validation of the software PRAEVAorta® 2 on 40 patients (principal objective).

The automatic measurements are compared to the physician measurements.

Procedure to follow:

Step 1. Inclusion and exclusion criteria validation Step 2. Demographic data and scanner references collection Step 3. CT scans (in DICOM format) collection Step 4. First Randomisation of the subjects' order Step 5. Determination of the measures by the physician with the standard method Step 6. Second randomisation of the subjects' order Step 7. Software analysis of the images with PRAEVAorta® Suite and Physician trust opinion In step 7, physicians will have to indicate if, based on the report generated by PRAEVAorta® 2, they trust the software measures or they do not, in order to validate clinical safety.

All data will be written in the e-CRF. The comparison of data will be done during the statistical analysis. The occurrence of device deficiencies will also be notified in the e-CRF.

A Mid-term report will be written by the end of part 1.

Part 2: Post-op follow-up of antero-posterior migration of stents and evaluation of the risk of endoleaks (secondary objective) The antero-posterior migration of stents will be analysed thanks to the software analysis.

This part is realised on post-op CT scan of 50 patients who have undergone a EVAR surgery. The 50 patients are composed of the 25 patients with an AAA, included in part 1 with 25 more in order to have more significant results.

Step 1. Inclusion and exclusion criteria validation for the 25 more patients Step 2. Demographic data and scanner references collection Step 3. CT scans (in DICOM format) collection Step 4. Software analysis of the images with PRAEVAorta® Suite All data will be written in the eCRF. The comparison of data will be done during the statistical analysis. The occurrence of device deficiencies will also be notified in the eCRF.

The final report will be written when both part of the study are realised.

Statistics:

Aggregated data analysed as treated and per subgroup. Descriptive analysis

* Pearson's coefficient correlation
* Absolute mean discrepancy per measurements
* Global mean and standard deviation per measurement endpoint
* Ratio for a measure
* Maximum aortic diameter ratio
* Computational analysis time The duration of the semi-automatic segmentation manually corrected by the 2 surgeons was reported and compared to the fully automatic method.
* Detectable and non-detectable error rate for safety evaluation
* Calculation of false positive, false negative, sensibility, specificity, positive predictive values, negative predictive values and likelihood ratio (LR+ and LR-). Inferential analysis Objective: comparing an observed proportion p1 with a theoretical proportion p0 p1: proportion of adequate data p0: theoretical proportion: 90% A one-sided right test will be realised to evaluate the comparison

Evaluation criteria:

Principal criteria:

• 90% of the patients shaw 90% of adequacy.

Secondary criteria:

Evaluation of the measurements and the segmentations:

* The mean discrepancy shall be ≤ 5mm
* Pearson correlation shall be ≥ 90%

Evaluation of risks:

* Unanticipated risks should not be critical Evaluation of the security
* The detectable error rate shall be ≥ 95%
* The non-detectable error rate shall be ≤ 5% Evaluation of PRAEVAorta® Web
* No critical bug No critical unanticipated risks

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Thoraco-abdominal Aneurysm
* Thoracic aortic aneurysm
* Or Infra-renal abdominal aortic aneurysm
* Or Juxta renal abdominal aortic aneurysm
* With or without calcification
* With or without stent

For part 2: patient treated by endurant (Medtronic) with sideways displacement during follow-up (more than 5mm)

Exclusion Criteria:

Patients with

* Ruptured aneurysms,
* Aortic dissections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with diagnosed or suspicion of an aortic aneurysm.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
orthogonal maximum diameter of the aorta (mm) | 3 months
Thoraco-Aortic lengths of the aorta (in mm) | 3 months
  * Proximal neck length
  * Infrarenal Aortic length
  * Left common Iliac artery length
  * Right common Iliac artery length
Infrarenal volume of the aorta (in cm3) | 3 months
  * Volume circulating
  * Intraluminal thrombus volume
  * Total volume
Aorta and iliacs diameters at several places (in mm) | 3 months
  * Aortic diameter above the uppermost renal artery
  * Upper proximal Neck Diameter
  * Neck Diameter 5mm under the lower renal
  * Neck Diameter 10mm under the lower renal
  * Neck Diameter 15mm under the lower renal
  * Neck diameter 20mm under the lower renal
  * Lower proximal Neck Diameter
  * Proximal right common Iliac artery Diameter
  * Middle right common iliac artery Diameter
  * Distal right common Iliac artery Diameter
  * Distal right external iliac artery Diameter
  * Proximal left common Iliac artery Diameter
  * Middle left common iliac artery Diameter
  * Distal left common iliac artery Diameter
  * Distal left external Iliac Diameter
  * Aortic bifurcation diameter
Suprarenal angulation (in hour and degree) | 3 months
  Angle between the suprarenal aorta and the neck
Infrarenal angulation (in hour and degree) | 3 months
  Angle between the neck and aneurysm

SECONDARY OUTCOMES:
Healthcare professional trust questionnaire | 2 days
  Do the professional trust or not the result returned by the software ? Yes or No reported in the CRF
Scan analyse time from segmentation to measurements | 3 months
  Time for analysis by the surgeon from segmentation to measurements Time for analysis by the automatique software from segmentation to measurement
Unanticipated risks | 3 days
  Risks that haven't been anticipated by Nurea, related to the use of the software
Number of male and female | 1 day
  the patient sex is collected in the CRF
Number of patient per age | 1 day
  the patient age is collected in the CRF

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Dr. SALOMON DU MONT, Principal Investigator — Centre Hospitalier Universitaire Jean Minjoz Besançon
Locations (1):
- Centre Hospitalier Universitaire Jean Minjoz, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moll FL, Powell JT, Fraedrich G, Verzini F, Haulon S, Waltham M, van Herwaarden JA, Holt PJ, van Keulen JW, Rantner B, Schlosser FJ, Setacci F, Ricco JB; European Society for Vascular Surgery. Management of abdominal aortic aneurysms clinical practice guidelines of the European society for vascular surgery. Eur J Vasc Endovasc Surg. 2011 Jan;41 Suppl 1:S1-S58. doi: 10.1016/j.ejvs.2010.09.011. No abstract available. PMID 21215940
- [Background] Szilagyi DE, Elliott JP, Smith RF. Clinical fate of the patient with asymptomatic abdominal aortic aneurysm and unfit for surgical treatment. Arch Surg. 1972 Apr;104(4):600-6. doi: 10.1001/archsurg.1972.04180040214036. No abstract available. PMID 5013802
- [Background] Scott RA, Wilson NM, Ashton HA, Kay DN. Influence of screening on the incidence of ruptured abdominal aortic aneurysm: 5-year results of a randomized controlled study. Br J Surg. 1995 Aug;82(8):1066-70. doi: 10.1002/bjs.1800820821. PMID 7648155
- [Background] Ashton HA, Buxton MJ, Day NE, Kim LG, Marteau TM, Scott RA, Thompson SG, Walker NM; Multicentre Aneurysm Screening Study Group. The Multicentre Aneurysm Screening Study (MASS) into the effect of abdominal aortic aneurysm screening on mortality in men: a randomised controlled trial. Lancet. 2002 Nov 16;360(9345):1531-9. doi: 10.1016/s0140-6736(02)11522-4. PMID 12443589
- [Background] Norman PE, Jamrozik K, Lawrence-Brown MM, Le MT, Spencer CA, Tuohy RJ, Parsons RW, Dickinson JA. Population based randomised controlled trial on impact of screening on mortality from abdominal aortic aneurysm. BMJ. 2004 Nov 27;329(7477):1259. doi: 10.1136/bmj.38272.478438.55. Epub 2004 Nov 15. PMID 15545293
- [Background] Powell JT, Brown LC, Forbes JF, Fowkes FG, Greenhalgh RM, Ruckley CV, Thompson SG. Final 12-year follow-up of surgery versus surveillance in the UK Small Aneurysm Trial. Br J Surg. 2007 Jun;94(6):702-8. doi: 10.1002/bjs.5778. PMID 17514693
- [Background] Lederle FA, Johnson GR, Wilson SE, Chute EP, Littooy FN, Bandyk D, Krupski WC, Barone GW, Acher CW, Ballard DJ. Prevalence and associations of abdominal aortic aneurysm detected through screening. Aneurysm Detection and Management (ADAM) Veterans Affairs Cooperative Study Group. Ann Intern Med. 1997 Mar 15;126(6):441-9. doi: 10.7326/0003-4819-126-6-199703150-00004. PMID 9072929
- [Background] Walker TG, Kalva SP, Yeddula K, Wicky S, Kundu S, Drescher P, d'Othee BJ, Rose SC, Cardella JF; Society of Interventional Radiology Standards of Practice Committee; Interventional Radiological Society of Europe; Canadian Interventional Radiology Association. Clinical practice guidelines for endovascular abdominal aortic aneurysm repair: written by the Standards of Practice Committee for the Society of Interventional Radiology and endorsed by the Cardiovascular and Interventional Radiological Society of Europe and the Canadian Interventional Radiology Association. J Vasc Interv Radiol. 2010 Nov;21(11):1632-55. doi: 10.1016/j.jvir.2010.07.008. Epub 2010 Sep 29. No abstract available. PMID 20884242
- [Background] Ghouri M, Krajcer Z. Endoluminal abdominal aortic aneurysm repair: the latest advances in prevention of distal endograft migration and type 1 endoleak. Tex Heart Inst J. 2010;37(1):19-24. PMID 20200623
- [Background] Tonnessen BH, Sternbergh WC 3rd, Money SR. Mid- and long-term device migration after endovascular abdominal aortic aneurysm repair: a comparison of AneuRx and Zenith endografts. J Vasc Surg. 2005 Sep;42(3):392-400; discussion 400-1. doi: 10.1016/j.jvs.2005.05.040. PMID 16171578
- [Background] Wyss TR, Brown LC, Powell JT, Greenhalgh RM. Rate and predictability of graft rupture after endovascular and open abdominal aortic aneurysm repair: data from the EVAR Trials. Ann Surg. 2010 Nov;252(5):805-12. doi: 10.1097/SLA.0b013e3181fcb44a. PMID 21037436
- [Background] Vorp DA, Vande Geest JP. Biomechanical determinants of abdominal aortic aneurysm rupture. Arterioscler Thromb Vasc Biol. 2005 Aug;25(8):1558-66. doi: 10.1161/01.ATV.0000174129.77391.55. PMID 16055757
- [Background] Nicholls SC, Gardner JB, Meissner MH, Johansen HK. Rupture in small abdominal aortic aneurysms. J Vasc Surg. 1998 Nov;28(5):884-8. doi: 10.1016/s0741-5214(98)70065-5. PMID 9808857
- [Background] Powell JT, Sweeting MJ, Brown LC, Gotensparre SM, Fowkes FG, Thompson SG. Systematic review and meta-analysis of growth rates of small abdominal aortic aneurysms. Br J Surg. 2011 May;98(5):609-18. doi: 10.1002/bjs.7465. Epub 2011 Mar 17. PMID 21412998
- [Background] Lindholt JS, Vammen S, Juul S, Henneberg EW, Fasting H. The validity of ultrasonographic scanning as screening method for abdominal aortic aneurysm. Eur J Vasc Endovasc Surg. 1999 Jun;17(6):472-5. doi: 10.1053/ejvs.1999.0835. PMID 10375481
- [Background] Long A, Rouet L, Lindholt JS, Allaire E. Measuring the maximum diameter of native abdominal aortic aneurysms: review and critical analysis. Eur J Vasc Endovasc Surg. 2012 May;43(5):515-24. doi: 10.1016/j.ejvs.2012.01.018. Epub 2012 Feb 14. PMID 22336051
- [Background] Ellis M, Powell JT, Greenhalgh RM. Limitations of ultrasonography in surveillance of small abdominal aortic aneurysms. Br J Surg. 1991 May;78(5):614-6. doi: 10.1002/bjs.1800780529. PMID 2059819
- [Background] Beales L, Wolstenhulme S, Evans JA, West R, Scott DJ. Reproducibility of ultrasound measurement of the abdominal aorta. Br J Surg. 2011 Nov;98(11):1517-25. doi: 10.1002/bjs.7628. Epub 2011 Aug 22. PMID 21861264
- [Background] Parr A, Jayaratne C, Buttner P, Golledge J. Comparison of volume and diameter measurement in assessing small abdominal aortic aneurysm expansion examined using computed tomographic angiography. Eur J Radiol. 2011 Jul;79(1):42-7. doi: 10.1016/j.ejrad.2009.12.018. Epub 2010 Jan 12. PMID 20061105
- [Background] Parr A, McCann M, Bradshaw B, Shahzad A, Buttner P, Golledge J. Thrombus volume is associated with cardiovascular events and aneurysm growth in patients who have abdominal aortic aneurysms. J Vasc Surg. 2011 Jan;53(1):28-35. doi: 10.1016/j.jvs.2010.08.013. PMID 20934838
- [Background] Stenbaek J, Kalin B, Swedenborg J. Growth of thrombus may be a better predictor of rupture than diameter in patients with abdominal aortic aneurysms. Eur J Vasc Endovasc Surg. 2000 Nov;20(5):466-9. doi: 10.1053/ejvs.2000.1217. PMID 11112467
- [Background] Houard X, Ollivier V, Louedec L, Michel JB, Back M. Differential inflammatory activity across human abdominal aortic aneurysms reveals neutrophil-derived leukotriene B4 as a major chemotactic factor released from the intraluminal thrombus. FASEB J. 2009 May;23(5):1376-83. doi: 10.1096/fj.08-116202. Epub 2009 Jan 9. PMID 19136615
- [Background] Houard X, Rouzet F, Touat Z, Philippe M, Dominguez M, Fontaine V, Sarda-Mantel L, Meulemans A, Le Guludec D, Meilhac O, Michel JB. Topology of the fibrinolytic system within the mural thrombus of human abdominal aortic aneurysms. J Pathol. 2007 May;212(1):20-8. doi: 10.1002/path.2148. PMID 17352452
- [Background] Satta J, Laara E, Juvonen T. Intraluminal thrombus predicts rupture of an abdominal aortic aneurysm. J Vasc Surg. 1996 Apr;23(4):737-9. doi: 10.1016/s0741-5214(96)80062-0. No abstract available. PMID 8627917
- [Background] Speelman L, Schurink GW, Bosboom EM, Buth J, Breeuwer M, van de Vosse FN, Jacobs MH. The mechanical role of thrombus on the growth rate of an abdominal aortic aneurysm. J Vasc Surg. 2010 Jan;51(1):19-26. doi: 10.1016/j.jvs.2009.08.075. Epub 2009 Nov 27. PMID 19944551
- [Background] Georgakarakos E, Ioannou CV, Kamarianakis Y, Papaharilaou Y, Kostas T, Manousaki E, Katsamouris AN. The role of geometric parameters in the prediction of abdominal aortic aneurysm wall stress. Eur J Vasc Endovasc Surg. 2010 Jan;39(1):42-8. doi: 10.1016/j.ejvs.2009.09.026. Epub 2009 Nov 10. PMID 19906549
- [Background] Kauffmann C, Tang A, Therasse E, Giroux MF, Elkouri S, Melanson P, Melanson B, Oliva VL, Soulez G. Measurements and detection of abdominal aortic aneurysm growth: Accuracy and reproducibility of a segmentation software. Eur J Radiol. 2012 Aug;81(8):1688-94. doi: 10.1016/j.ejrad.2011.04.044. Epub 2011 May 20. PMID 21601403
- [Background] Wever JJ, Blankensteijn JD, Th M Mali WP, Eikelboom BC. Maximal aneurysm diameter follow-up is inadequate after endovascular abdominal aortic aneurysm repair. Eur J Vasc Endovasc Surg. 2000 Aug;20(2):177-82. doi: 10.1053/ejvs.1999.1051. PMID 10942691
- [Background] Kritpracha B, Beebe HG, Comerota AJ. Aortic diameter is an insensitive measurement of early aneurysm expansion after endografting. J Endovasc Ther. 2004 Apr;11(2):184-90. doi: 10.1583/03-976.1. PMID 15056034
- [Background] van Keulen JW, van Prehn J, Prokop M, Moll FL, van Herwaarden JA. Potential value of aneurysm sac volume measurements in addition to diameter measurements after endovascular aneurysm repair. J Endovasc Ther. 2009 Aug;16(4):506-13. doi: 10.1583/09-2690.1. PMID 19702341
- [Background] Bley TA, Chase PJ, Reeder SB, Francois CJ, Shinki K, Tefera G, Ranallo FN, Grist TM, Pozniak M. Endovascular abdominal aortic aneurysm repair: nonenhanced volumetric CT for follow-up. Radiology. 2009 Oct;253(1):253-62. doi: 10.1148/radiol.2531082093. Epub 2009 Jul 31. PMID 19703867
- [Background] Nambi P, Sengupta R, Krajcer Z, Muthupillai R, Strickman N, Cheong BY. Non-contrast computed tomography is comparable to contrast-enhanced computed tomography for aortic volume analysis after endovascular abdominal aortic aneurysm repair. Eur J Vasc Endovasc Surg. 2011 Apr;41(4):460-6. doi: 10.1016/j.ejvs.2010.11.027. Epub 2010 Dec 31. PMID 21195639
- [Background] Prinssen M, Verhoeven EL, Verhagen HJ, Blankensteijn JD. Decision-making in follow-up after endovascular aneurysm repair based on diameter and volume measurements: a blinded comparison. Eur J Vasc Endovasc Surg. 2003 Aug;26(2):184-7. doi: 10.1053/ejvs.2002.1892. PMID 12917836
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Riambau V, Bockler D, Brunkwall J, Cao P, Chiesa R, Coppi G, Czerny M, Fraedrich G, Haulon S, Jacobs MJ, Lachat ML, Moll FL, Setacci C, Taylor PR, Thompson M, Trimarchi S, Verhagen HJ, Verhoeven EL, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus ES, Hinchliffe RJ, Kakkos S, Koncar I, Lindholt JS, Vega de Ceniga M, Vermassen F, Verzini F, Document Reviewers, Kolh P, Black JH 3rd, Busund R, Bjorck M, Dake M, Dick F, Eggebrecht H, Evangelista A, Grabenwoger M, Milner R, Naylor AR, Ricco JB, Rousseau H, Schmidli J. Editor's Choice - Management of Descending Thoracic Aorta Diseases: Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2017 Jan;53(1):4-52. doi: 10.1016/j.ejvs.2016.06.005. No abstract available. PMID 28081802
- [Background] Scott SW, Batchelder AJ, Kirkbride D, Naylor AR, Thompson JP. Late Survival in Nonoperated Patients with Infrarenal Abdominal Aortic Aneurysm. Eur J Vasc Endovasc Surg. 2016 Oct;52(4):444-449. doi: 10.1016/j.ejvs.2016.05.008. Epub 2016 Jun 30. PMID 27374814
- [Background] Claridge R, Arnold S, Morrison N, van Rij AM. Measuring abdominal aortic diameters in routine abdominal computed tomography scans and implications for abdominal aortic aneurysm screening. J Vasc Surg. 2017 Jun;65(6):1637-1642. doi: 10.1016/j.jvs.2016.11.044. Epub 2017 Feb 16. PMID 28216357
- [Background] Mell MW, Hlatky MA, Shreibati JB, Dalman RL, Baker LC. Late diagnosis of abdominal aortic aneurysms substantiates underutilization of abdominal aortic aneurysm screening for Medicare beneficiaries. J Vasc Surg. 2013 Jun;57(6):1519-23, 1523.e1. doi: 10.1016/j.jvs.2012.12.034. Epub 2013 Feb 12. PMID 23414696
- [Background] de Bruijne M, van Ginneken B, Viergever MA, Niessen WJ. Interactive segmentation of abdominal aortic aneurysms in CTA images. Med Image Anal. 2004 Jun;8(2):127-38. doi: 10.1016/j.media.2004.01.001. PMID 15063862
- [Background] Lopez-Linares K, Aranjuelo N, Kabongo L, Maclair G, Lete N, Ceresa M, Garcia-Familiar A, Macia I, Gonzalez Ballester MA. Fully automatic detection and segmentation of abdominal aortic thrombus in post-operative CTA images using Deep Convolutional Neural Networks. Med Image Anal. 2018 May;46:202-214. doi: 10.1016/j.media.2018.03.010. Epub 2018 Mar 27. PMID 29609054
- [Background] Ahmed S, Zimmerman SL, Johnson PT, Lai H, Kawamoto S, Horton KM, Fishman EK. MDCT interpretation of the ascending aorta with semiautomated measurement software: improved reproducibility compared with manual techniques. J Cardiovasc Comput Tomogr. 2014 Mar-Apr;8(2):108-14. doi: 10.1016/j.jcct.2013.12.009. Epub 2014 Jan 11. PMID 24568947
- [Background] Singh K, Jacobsen BK, Solberg S, Bonaa KH, Kumar S, Bajic R, Arnesen E. Intra- and interobserver variability in the measurements of abdominal aortic and common iliac artery diameter with computed tomography. The Tromso study. Eur J Vasc Endovasc Surg. 2003 May;25(5):399-407. doi: 10.1053/ejvs.2002.1856. PMID 12713777
- [Background] Caradu C, Spampinato B, Vrancianu AM, Berard X, Ducasse E. Fully automatic volume segmentation of infrarenal abdominal aortic aneurysm computed tomography images with deep learning approaches versus physician controlled manual segmentation. J Vasc Surg. 2021 Jul;74(1):246-256.e6. doi: 10.1016/j.jvs.2020.11.036. Epub 2020 Dec 9. PMID 33309556
- [Background] Taha AA, Hanbury A. Metrics for evaluating 3D medical image segmentation: analysis, selection, and tool. BMC Med Imaging. 2015 Aug 12;15:29. doi: 10.1186/s12880-015-0068-x. PMID 26263899
- [Background] Jongkind V, Yeung KK, Akkersdijk GJ, Heidsieck D, Reitsma JB, Tangelder GJ, Wisselink W. Juxtarenal aortic aneurysm repair. J Vasc Surg. 2010 Sep;52(3):760-7. doi: 10.1016/j.jvs.2010.01.049. Epub 2010 Apr 10. PMID 20382492